CLINICAL TRIAL: NCT01038544
Title: Endobronchial Ultrasound (EBUS) for Nodal Staging in Esophageal Cancer
Acronym: CT0003
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: C.E.T.O.C. - CHUM Endoscopic Tracheobronchial and Oesophageal Center (Unknown); Marcel and Rolande Gosselin Chair in Thoracic Surgical Oncology (Unknown); Fonds de la Recherche en Santé du Québec (Other Government); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CE 09.146
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2011-11

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Mediastinal lymph nodes; Staging; EBUS; EUS; Endobronchial Ultrasound; Endoscopic Ultrasound
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endoscopic Ultrasound (EUS) — Minimally Invasive Echo-Endoscopic Lymph Node Evaluation and Biopsy
  Other Names: minimally invasive mediastinal staging
Procedure: Endobronchial Ultrasound (EBUS) — Minimally Invasive Echo-Bronchoscopic Lymph Node Evaluation and Biopsy
  Other Names: minimally invasive mediastinal staging

SUMMARY:
The purpose of this study is determine if performing endobronchial ultrasound (EBUS) in addition to standard endoscopic ultrasound (EUS) can increase the precision and accuracy of staging esophageal cancer in comparison to EUS alone. The expectation is that EBUS can be used to biopsy lymph nodes that: (1) because of their position in the mediastinum would be inaccessible to EUS, or (2) would be inaccessible due to their position behind the esophageal tumor.

DETAILED DESCRIPTION:
1. Problem:

   Endoscopic ultrasound techniques are becoming more and more popular. The safety of these technologies has been demonstrated on multiple occasions. These minimally invasive trans-luminal techniques do not require general anesthesia and can be performed, rapidly, accurately and at low cost. Endobronchial ultrasound (EBUS) has been used by pulmonologists and thoracic surgeons primarily for the staging, diagnosis and management of lung cancer. Its efficacy and safety has been demonstrated in multiple studies.

   EBUS is not currently utilized by most centers in the staging of esophageal cancer. To date, no study has explored the possible use of EBUS for peritumoral lymph node biopsy, nor for biopsy of any suspicious mediastinal lymph nodes, not accessible by EUS. At Notre Dame Hospital, Centre Hospitalier de L'Universite de Montreal, all patients diagnosed with esophageal cancer undergo complete EUS staging followed by EBUS during the same procedure, in order to examine all the lymph nodes near or far from the primary tumor amenable to EBUS guided trans-bronchial biopsy. This is important because it allows physicians to bypass the primary tumor and pass through the normal (non-cancerous) bronchial wall, eliminating any chances of tumoral contamination of the sample. In addition, this also provides a much more complete mediastinal staging as it allows biopsy of a population of lymph nodes non-accessible to EUS biopsy. Thus far, we have performed EBUS in six patients with esophageal cancer with upstaging of the N stage of the tumor in two of these patients (33%). There have been no morbidities and all patients have been discharged home on the day of the procedure. EBUS was therefore able to change the treatment strategy, without adding any morbidity, discomfort or additional procedural time for two out of six patients.

   The proposed project will be the first study ever to evaluate the impact of EBUS on esophageal cancer staging as well as on the choice of therapy. This study consists of a prospective cohort study with no placebo group, all patients will have EBUS and stages obtained with and without EBUS will be compared as well as changes to the treatment plan based on EBUS staging.
2. Objectives:

   * Examine the impact of adding EBUS to the gold standard work-up on esophageal cancer staging.
   * Examine the impact of adding EBUS to the gold standard work-up on the treatment plan for patients newly diagnosed with esophageal cancer.
3. Methodology:

   The study consists of a prospective cohort study. Each patient will serve as his/her own control. All patients currently undergoing esophageal cancer staging in the Division of Thoracic Surgery at the CHUM will be approached for enrolment into the study.

   EUS followed by EBUS will be performed during the EUS staging procedure. The order of procedures for all patients is as follows: (1) Flexible Esophagoscopy with endoluminal biopsy, (2) Radial EUS for T staging (3) Linear EUS for lymph node biopsy and N staging, (4) Flexible Bronchoscopy for evaluation of the left mainstem bronchus for tumor invasion, (5) Linear EBUS for trans-tracheal and trans-bronchial lymph node biopsy.

   All FNA samples will be evaluated using standard methods by cytopathologists at the CHUM. Results will be evaluated for: (A) positivity, (B) negativity (no tumor cells, positive lymphocytes), (C) inadequacy (no tumor cells, no lymphocytes). A minimum of two passes will be performed into each lymph node.

   Patients will be discharged on the same day, as their procedure. Results will be discussed with them in a follow-up clinic appointment with their thoracic surgeon within 3 weeks of the procedure. Any procedure-related morbidity will be documented in the post-procedural period as well as at their follow-up appointment.
4. Expected Results:

We believe that by adding EBUS to the gold standard work up and staging of esophageal cancer, we can make a significant difference in esophageal cancer staging. This may also significantly change the choice of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven esophageal cancer
* Endoluminal esophageal mass without previous biopsy
* Medical suitability for endoscopic procedure
* Ability to consent

Exclusion Criteria:

* Patient on Coumadin (Warfarin) or Plavix (Clopidogrel) with inability to stop medication for 5 days prior to procedure
* Anatomy precluding EBUS
* Endobronchial tumor
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the accuracy of the combination of EUS and EBUS to correctly diagnose the presence or absence of mediastinal lymph node metastases compared to EUS alone. | 6 months intervals

SECONDARY OUTCOMES:
The safety of all diagnostic techniques will be evaluated and compared between techniques. | 6 months
Procedure-related morbidity | 6 months
Change in treatment plan based on EBUS | Study termination

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada